CLINICAL TRIAL: NCT06622616
Title: NUTRITIONAL INTERVENTION STUDY to EVALUATE the EFFECT of ACHETA DOMESTICUS POWDER CONSUMPTION on GLUCOSE HOMEOSTASIS and INTESTINAL DYSBIOSIS in HEALTHY and PREDIABETIC POPULATION
Acronym: DIBAN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: María Isabel Espinosa (Other)
Collaborators: Biomedical Research Institute Sols-Morreale (CSIC-UAM) (Unknown); Centro de BiologÃ-a Molecular Severo Ochoa, Spain (CBMSO) (Unknown); Epidisease S.L (Other); NUTRINSECT (Unknown)
Responsible Party: Sponsor-Investigator, María Isabel Espinosa, PhD, IMDEA Food
Organization: IMDEA Food (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMDEA FOOD; HORIZON-EIC-2023-PATHFINDER (Other Grant/Funding Number: EUROPEAN COMISION)
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Insulin Resistance; Type 2 Diabetes Mellitus with Features of Insulin Resistance
Keywords: Acheta Domesticus; Insect powder; Insulin resistance; microbiota; Artificial Inteligence
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: A pilot nutritional intervention study will be conducted that will be longitudinal, prospective, double-blind, randomized and parallel.
  The study will have two arms, the functional group with A. domesticus powder (n=60) and a placebo group that will take a vegetable protein powder with a similar macronutrient composition (n=60). This population will be classified according to sex and BMI, and their nutritional-metabolic status (insulin resistance or not).
Who Masked: Participant, Investigator
Masking Description: The study will be masked by using identical packaging for both the study group and the control group (placebo), which participants will consume at home or at the place where they eat, during the 12 weeks of the intervention. The packaging of the products will be carried out by the company supplying A. domesticus powder, Nutrinsect SRL (Italy), which is authorised to produce A. domesticus powder according to EFSA approval.
  The researchers will administer the product (with identical external appearance for both groups) individually to each participant.
  The randomisation will be carried out blindly, so that each of the participants and the researcher will not know which group (study or control) they have received. For this purpose, the product under study will be labeled with the protocol code and the letters A or B (or batch number) that will correspond to the functional and/or control product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Experimental): Los participantes consumirán 2 porciones de producto con polvo de A. domesticus (15 g. cada una) que podrán consumir al gusto en diferentes recetas. El producto estará incluido dentro de un plan de alimentación saludable normoproteico. Se les recomendará continuar con su actividad física habitual durante las 12 semanas de duración del estudio.
  Interventions: Dietary Supplement: EVALUATE THE EFFECT OF ACHETA DOMESTICUS POWDER CONSUMPTION ON GLUCOSE HOMEOSTASIS AND INTESTINAL DYSBIOSIS
- Control Group (Placebo Comparator): Participants will consume 2 portions of a product with a nutritional value similar to the study product, one at breakfast and one at dinner. The product will be included in a healthy, normoprotein diet plan. They will be advised to continue their usual physical activity during the 12 weeks of the study.
  Interventions: Dietary Supplement: EVALUATE THE EFFECT OF ACHETA DOMESTICUS POWDER CONSUMPTION ON GLUCOSE HOMEOSTASIS AND INTESTINAL DYSBIOSIS

INTERVENTIONS:
Dietary Supplement: EVALUATE THE EFFECT OF ACHETA DOMESTICUS POWDER CONSUMPTION ON GLUCOSE HOMEOSTASIS AND INTESTINAL DYSBIOSIS — The study will have two arms, the functional group with A. domesticus powder (n=60) and a placebo group that will take a vegetable protein powder with a similar macronutrient composition (n=60). This population will be classified according to sex and BMI, and their nutritional-metabolic status (insulin resistance or not).
  The study will include analysis of phenotypic data collection (medical history, lifestyle, diet, etc.); biochemical data: glucose, lipid, iron profile, blood count, and analysis of inflammation markers; genotyping, epigenetic analysis (methylation and mi-RNAs), targeted metabolomics (glycome and tryptophan) and metagenomic analysis of stool (16s rRNA sequencing for taxonomic identification study). Using continuous monitoring devices (glucose monitoring using a sensor and physical activity using an activity bracelet), lifestyle parameters (physical activity, circadian rhythms, sleep, stress, etc.) and blood glucose will be evaluated.

SUMMARY:
A nutritional intervention study is proposed to evaluate the association between the consumption of A. domesticus (insect protein) powder and the effect on insulin resistance and the microbiome, in order to generate personalized nutrition strategies through its analysis with artificial intelligence.

This study is expected to involve 120 healthy volunteers between 18 and 65 years old, with or without insulin resistance, who will be recruited by IMDEA-Food. This is a 12-week nutritional intervention study, so you must come to Institute IMDEA-Food for a first screening visit (V0) and, if you meet the study inclusion criteria and are still interested in volunteering for the study, you will be informed about the study, sign the informed consent form and be scheduled for 2 more visits (V1 or initial zero-time, and V2 or final) at IMDEA-Food's facilities.

DETAILED DESCRIPTION:
In visit 1 (basal visit), the participant will provide a stool sample (for microbiota analysis), a fasting blood sample (for biochemical, genetic, epigenetic and metabolomic analysis) and then go to the nutrition consultation where medical history data and lifestyle habits will be collected, a nutritional assessment will be made and the completed questionnaires will be corrected. In addition, they will be provided with continuous glucose monitoring sensors and an activity wristband to record lifestyle patterns. The glucose sensors will be used for the first 14 and last 14 days of the intervention. In addition, all participants will be provided with the required amount of product until the next visit, as well as how to consume, store, and ideas for consumption. In addition, a balanced (normoprotein) and varied diet and physical activity guidelines will be explained.

In the second visit (final), the participant will again submit a stool sample (for microbiota analysis), a fasting blood sample will be taken (for biochemical, epigenetic and metabolomic analysis) and then they will go to the nutrition clinic where a nutritional assessment will be made and the completed questionnaires will be corrected. In addition, the glucose sensor and the activity bracelet will be removed.

During the intervention phase of the study, participants will be able to come to the center for the collection of more product as well as for the review and troubleshooting of any problems with the sensors that may arise. In turn, halfway through the study (6 weeks), a telephone survey will be conducted to participants to avoid travel, in order to assess the degree of adherence and possible adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 65 years of age.
* Adequate cultural level and understanding of the clinical study.
* Agree to participate voluntarily in the study and give their informed consent in writing.

Exclusion Criteria:

* Subjects with dementia, mental illness or decreased cognitive function that prevents understanding of the study.
* Subjects with celiac disease or serious diseases (tumour, immunological, intestinal, metabolic, cardiovascular processes, etc.).
* BMI < 18 or ≥ 35.
* Pregnant or breastfeeding women.
* Being a socially vulnerable person.
* Subjects whit chronic pharmacological treatment for weight loss, insulin or antibiotic treatment in the month prior to the start of the intervention or during it.
* Subjects with food allergies, especially to mollusks and their by-products, dust mites, chickpeas or soy (the product may contain traces of soy and gluten).

  * Subjects who refuse to be monitored by sensors, collect samples, draw blood and nutritional visits.
  * Subjects who reject the consumption of products made with alternative proteins (insect powder).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
insulin resistance (HOMA) | 3 months
  The primary endpoint will be changes in insulin resistance values after 3 months of intervention.

IPD SHARING:
Plan to Share IPD: Undecided